CLINICAL TRIAL: NCT06754527
Title: Emotion Regulation Intervention to Prevent Substance Use Among Youth in the Child Welfare System
Brief Title: Options for Navigating Talking About Risk and Adolescent Choices
Acronym: ON-TRAC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ON-TRAC (unknown Protocol ID); R61DA059785 (NIH)
Record Dates: First submitted 2024-12-23; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Substance Use (Drugs, Alcohol); Substance Use Risk; Substance Use; Emotion Regulation; Risk Reduction Behavior; Risk Reduction
Keywords: adolescent substance use; emotion regulation; risk reduction
MeSH Terms: conditions — Substance-Related Disorders; Emotional Regulation; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ON-TRAC Intervention (Experimental): Web-based emotion regulation and substance use intervention
  Interventions: Behavioral: ON-TRAC
- Waitlist Control (No Intervention): Control participants are assessed on the same schedule as the treatment condition and offered the intervention after the 8-month follow-up

INTERVENTIONS:
Behavioral: ON-TRAC — Online tablet-based intervention that teaches youth emotion regulation skills and integrates substance use prevention content
  Arms: ON-TRAC Intervention

SUMMARY:
This study will examine the effectiveness of ON-TRAC (Options for Navigating Talking about Risk and Adolescent Choices), which is an online substance use prevention program that also teaches emotion regulation skills. 200 adolescents, 12-15 years of age, will be randomized to ON-TRAC or a wait list comparison group (who will be offered the intervention at the end of their study participation) to determine impact on substance use, emotion regulation abilities, mental health symptoms, and other risk behavior outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Contact with the Rhode Island child welfare system
* Caregiver who is a parent/guardian of a child who experienced maltreatment
* Caregiver who speaks English or Spanish
* Caregiver who does not have developmental delays
* Adolescent who is between 12-15 years of age
* Adolescent who is fluent in English
* Adolescent who has active follow-up with the Rhode Island child welfare system due to an indicated finding of abuse or neglect in the past year

Exclusion Criteria:

* Adolescent who cannot read at a 4th grade level
* Adolescent who has a sibling who has participated in the program
* Adolescent who has developmental delays
* Adolescent who lacks parental consent for the study

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Timeline Follow Back | Baseline, 2-, 5-, and 8-months
  A calendar assisted daily substance use estimation method obtained by interview. Days used will serve as primary outcome. More days used represent more substance use.

SECONDARY OUTCOMES:
Drinking Refusal Self-Efficacy Questionnaire - Shortened Adolescent Version | Baseline, 2-, 5-, and 8-months
  Assesses self-efficacy to resist alcohol use. Scores range from 9 to 54. Higher scores represent greater drinking refusal self-efficacy.
Drinking Refusal Self-Efficacy Questionnaire - Shortened Adolescent Version (Adapted for Marijuana Use) | Baseline, 2-, 5-, and 8-months
  Assesses self-efficacy to resist marijuana use. Scores range from 9 to 54. Higher scores represent greater marijuana refusal self-efficacy.

OTHER OUTCOMES:
Youth Risk Behavior Surveillance Survey | Baseline, 2-, 5-, and 8-months
  Single items assess other risk behaviors such as sexual risk or violence behaviors. Endorsement of each individual item indicates engagement in the risk behavior.
Patient-Reported Outcome Measures Information System - Anger Scale | Baseline, 2-, 5-, and 8-months
  Assesses symptoms of mental health and social functioning. Scores range from 5 to 25. Higher scores indicate greater anger.
Difficulties in Emotion Regulation Scale | Baseline, 2-, 5-, and 8-months
  Assesses perceptions of emotion regulation skills. Scores range from 18-90. Higher scores indicate more difficulty regulating emotions.
Emotion Regulation Behaviors Scale | Baseline, 2-, 5-, and 8-months
  Assesses use of emotion regulation behaviors taught in the intervention. Scores range from 9 to 36. Higher scores indicate more frequent use of the strategies taught.
Diagnostic Analysis of Nonverbal Accuracy-2 | Baseline, 2-, and 8-months
  Computer-based measure that asks participants to identify the emotion of facial expressions displayed in photographs. Scores range from 0 to 20. Higher scores indicate better identification of emotions.
Behavioral Indicator of Resiliency to Distress | Baseline, 2-, and 8-months
  Computerized frustration task in which participants are given the option to quit at any time. Scores range from 0 to 300 seconds. Higher scores indicate more persistence in a frustrating task.
Self-Efficacy Questionnaire for Children | Baseline, 2-, 5-, and 8-months
  Assesses perception of ability to cope with negative emotions. Scores range from 8 to 40. Higher scores indicate greater perceived ability to cope with negative emotions.
Implicit Theories of Emotions for Children - Self subscale | Baseline, 2-, 5-, and 8-months
  Assesses beliefs about the controllability of emotions. Scores range from 6 to 36. Higher scores indicate stronger beliefs about the controllability of emotions.
Respiratory sinus arrhythmia | Baseline and 2-month follow up
  Collected in response to virtual reality scenes, RSA is a physiological marker of emotion regulation processes calculated from heart rate variability as an index of parasympathetic activity.
Feasibility and Acceptability Scale | 2-month follow-up (ON-TRAC group only)
  Assesses acceptability of digital interventions to assess implementation outcomes. Scores range from 5 to 25. Higher scores indicate greater acceptability of the intervention.
System Usability Scale | 2-month follow-up (ON-TRAC group only)
  Assesses usability of technology programs to assess implementation outcomes. Scores range from 10 to 50. Higher scores indicate greater usability of the intervention.